CLINICAL TRIAL: NCT01142336
Title: Effects of Simvastatin on CSF AD Biomarkers in Cognitively Normal Subjects
Brief Title: Effects of Simvastatin on Biomarkers
Acronym: SimBio
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Institute for Biomedical and Clinical Research (Other); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gail Li, Associate Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 37373; 00183 (Other: VA Puget Sound Health System MIRB#)
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Prevention; Spinal Fluid; Biomarkers; Simvastatin
MeSH Terms: conditions — Alzheimer Disease | interventions — Simvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Simvastatin (Experimental): Simvastatin 40mg qHS for 1 year
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo 1 tablet qHS for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40mg qHS for 1 year
  Other Names: Zocor
  Arms: Simvastatin
Drug: Placebo — Placebo 1 tablet qHS for 1 year
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
A year-long randomized, double-blind, placebo-controlled trial of simvastatin to see if it produces beneficial changes in cerebral spinal fluid proteins associated with Alzheimer's disease.

DETAILED DESCRIPTION:
The purpose of this study is to see if a drug called simvastatin (brand name Zocor) beneficially affects the level of certain molecules (such as proteins) in the spinal fluid of people. The molecules the investigators are measuring are thought to be important in the development of Alzheimer's disease (AD), and the investigators are testing whether simvastatin can change proteins to a level that is associated with a reduced risk for AD.

Simvastatin has been approved by the United States Food and Drug Administration (FDA) for the treatment of high cholesterol and to reduce the risk of coronary artery disease. It is an investigational drug in this study.

Participants will be randomly assigned to Placebo or Simvastatin. The investigators and the participant will be blinded. Randomization will be stratified by age and gender.

This study is being funded by the National Institute on Aging. The investigators will take part in this study at the VA Puget Sound Health Care System.

This study will last up to 1 year. Participants will be asked to come to the VA in Seattle a total of 9 times, 2 of those times will be for lumbar punctures (also known as a spinal tap).

The investigators would also like to ask a person who knows the participant well (such as a spouse, child, sibling, or good friend) some questions about the participant's health, memory, mood and behavior, and abilities to do daily tasks at the beginning and the end of the study.

Participants must be cognitively normal, healthy, willing to have a lumbar puncture, and not need or take any medications to control cholesterol.

ELIGIBILITY:
Inclusion Criteria (participants must meet the following criteria)

* If female of childbearing potential, must have negative pregnancy test at baseline, and all subsequent visits.
* Age 45 to 64 years inclusive.
* Considered cognitively normal with no evidence of memory or other cognitive impairments (MMSE >26, Logical Memory delayed recall > 6, CDR score of 0).
* Normal or only mildly elevated cholesterol which does not require drug therapy based on National Cholesterol Education Program Adult Treatment Panel III (NCEP/ATP-III) guidelines.
* An LDL level above 70mg/dL.
* Hamilton Depression Scale (HAM-D) score < 12.
* BMI between 18 - 34 (or exception made by MD).
* In good recent general health (i.e., no trauma or infection in the 4 weeks before LP).
* On stable dose of non-exclusionary medications for the 4 weeks preceding the LP.
* Platelet count >100,000.

Exclusion Criteria (participants must NOT satisfy any of the following conditions)

* Any contraindications to LP, such as spinal deformity, severe disease or infection in the LP region, bleeding tendency, anticoagulant or blood-thinning medications.
* Taken a statin medication in the past 12 months.
* Any clinically significant laboratory abnormalities.
* Any neurological disorders: multiple sclerosis, epilepsy, stroke, Parkinson's, other degenerative CNS disorders, or neuropathy with radicular involvement.
* Acute or chronic major psychiatric disorders: schizophrenia, affective disorders, or severe anxiety disorders. (Dysthymia allowed, history of MDD allowed if currently in remission)
* Unstable or poorly controlled medical problems such as: heart failure, diabetes (poorly controlled or insulin dependent), hypertension (BP >160/100), pulmonary disease with hypoxia or hypercapnia, significant liver disease or known hepatitis C seropositivity, renal failure, treatment for cancer in the past 2 years (other than non-melanoma skin cancer) or known HIV positive status.
* Use of illegal drugs or alcohol abuse (>2 drinks/day or 10/week) within the past year.
* Concurrent participation in another investigational drug study.
* Use of any exclusionary medications in the 4 weeks prior to screening:

  * Drugs which could interact with statins: itraconazole, ketoconazole, erythromycin, clarithromycin, HIV protease inhibitors, nefazodone, amiodarone, cyclosporine, isoniazid, quinidine, or large quantities of grapefruit juice (>1 quart daily)
  * Central nervous system acting medications: antipsychotics, anti-Parkinson's disease medications, anti convulsants, or CNS stimulants
  * Chronic use of benzodiazepines, sedating antihistamines, or other sedative-hypnotic agents (prn use is allowed as long as it is not within 72 hours of LP or cognitive testing)
  * Medications affecting coagulation and/or inflammation: coumadin, potent anti-inflammatory medications (hydrocortisone, methotrexate or other potent immune-modulating medications), and anti-HIV medications (Aspirin up to 325 mg/day is allowed.)
  * Lipid-lowering drugs: fibrates or niacin >500mg/day (stable dose of omega-3 is allowed)
* Does the subject's family history meet any of the following criteria?

  * Both parents had/have dementia
  * On one side of the family, over two consecutive generations three relatives had/have dementia?
  * One parent had an onset of dementia before age 60?
* Does the subject have a major active autoimmune or immunological disorder?

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Li, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Statin-naïve middle-aged adults were recruited for this single-site trial (Seattle, WA) from the University of Washington Alzheimer's Disease Research Center Registry or the community through newsletters, websites, educational talks, health fairs, local clinics, and newspaper and magazine advertisements.
Pre-assignment Details: 917 people were pre-screened by phone for eligibility, 400 did not respond or declined, 457 did not meet inclusion/exclusion criteria.
  60 completed a full screen visit. Of these 60 potential participants, 2 were lost to follow-up after screen, 2 withdrew, 7 screen failed and 49 were enrolled and randomized.
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 26 | 23
Completed | 25 | 21
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Simvastatin | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (4.9) | 55.7 (4.5) | 55.9 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49
CSF Aβ42 level [Mean (Standard Deviation); unit: pg/ml] | 515 (113) | 520 (114) | 517 (113)
CSF total tau level [Mean (Standard Deviation); unit: pg/ml] | 43 (17) | 38 (16) | 41 (16)
CSF ptau level [Mean (Standard Deviation); unit: pg/ml] | 31 (15) | 27 (10) | 29 (12)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aβ42 in Cerebrospinal Fluid (CSF) at 1 Year
Description: CSF Aβ42 concentration were measured at baseline and after 1-year intervention.
Time Frame: 1-year change of CSF Aβ42 from baseline
Population: In the Placebo group, 1 participant was dropped due to AE and 1 was lost to follow-up.
  In the Simvastatin group, 1 participant was dropped due to AE. These 3 participants were not included in the primary analysis per analysis plan.
  All these 3 subjects were not included in the primary analysis based on our per protocol analysis plan.
Measure: Mean (Standard Deviation); unit: 1-yr change, pg/ml
Groups:
- Placebo: 1 tab qHS for 1 year
- Simvastatin: 40mg qHS for 1 year
Arm/Group | Placebo | Simvastatin
Number analyzed (Participants) | 21 | 25
1-yr change, pg/ml | 5.3 (31) | 0.5 (42)
Statistical Analysis 1: Comparison: Placebo vs Simvastatin; Test type: Superiority; p = 0.53, ANCOVA — Threshold for significance: 0.05, adjust for 3 primary outcomes using Holm Correction; Response variable was Aβ42 in CSF at 1 year, and predictor variables were Aβ42 in CSF at baseline, treatment group, age, sex, and APOE e4 allele

2. Primary Outcome: Change From Baseline in CSF Total Tau at 1 Year
Description: CSF total tau was measured at baseline and after 1-year of intervention
Time Frame: 1-yr change
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Placebo: 1 tablet qHS for 1 year
Arm/Group | Placebo | Simvastatin
Number analyzed (Participants) | 21 | 25
pg/ml | -0.1 (3.9) | 1.6 (4.7)
Statistical Analysis 1: Comparison: Placebo vs Simvastatin; Test type: Superiority; p = 0.36, ANCOVA — Threshold for significance: 0.05, adjusted for 3 primary outcomes using Holm correction; Response variable was total tau in CSF at 1 year, and predictor were total tau in at baseline, treatment group, age, sex, and APOE e4 allele status

3. Primary Outcome: Change From Baseline in CSF ptau181 at 1 Year
Description: ptau 181 measured in CSF at baseline and after 1-year intervention
Time Frame: 1-year change from baseline
Measure: Mean (Standard Deviation); unit: 1-yr change (final - baseline), pg/ml
Arm/Group | Placebo | Simvastatin
Number analyzed (Participants) | 21 | 25
1-yr change (final - baseline), pg/ml | -2.9 (12.9) | 1.7 (6.3)
Statistical Analysis 1: Comparison: Placebo vs Simvastatin; Test type: Superiority; p = 0.25, ANCOVA — Threshold for significance: 0.05, adjusted for 3 primary outcomes using Holm correction; Response variable was p-tau181 in CSF at 1 year, and predictor were p-tau181 in at baseline, treatment group, age, sex, and APOE e4 allele status

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event information was collected systematically at phone and in-person safety visits spaced 6 weeks to 3 months apart for the duration of the 1 year study.
Arm/Group | Simvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 26/26 | 22/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin (N=26) | Placebo (N=23)
Headache (General disorders) | 7 | 8 — New or worsening Headache
Nausea (Gastrointestinal disorders) | 3 | 2 — New or worsening Nausea
Diarrhea (Gastrointestinal disorders) | 5 | 2 — New or worsening diarrhea
Constipation (Gastrointestinal disorders) | 3 | 2 — New or worsening constipation
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 14 | 9 — New or worsening upper respiratory infection
Memory Problems (Psychiatric disorders) | 1 | 5 — Self-reported new or worsening memory problems
Depressed Mood (Psychiatric disorders) | 2 | 4 — Self-reported new or worsening depressed mood
Anxiety (Psychiatric disorders) | 3 | 8 — Self-reported new or worsening anxiety
Insomnia (General disorders) | 7 | 5 — New or worsening insomnia
Muscle Pain (Musculoskeletal and connective tissue disorders) | 6 | 8 — New or worsening muscle pain
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 — New or worsening muscle weakness
Elevated Blood Glucose (Metabolism and nutrition disorders) | 3 | 5 — Fasting Blood Glucose lab reading above normal limits
Elevated serum glutamic-oxaloacetic transaminase (SGOT) (Hepatobiliary disorders) | 3 | 5 — SGOT lab reading above normal limits
Elevated Serum glutamic pyruvic transaminase (SGPT) (Hepatobiliary disorders) | 6 | 1 — SGPT lab reading above normal limits
Elevated serum creatine phosphokinase (CPK) (Musculoskeletal and connective tissue disorders) | 7 | 6 — serum CPK lab reading above normal limits

LIMITATIONS AND CAVEATS:
Sample size is small and statistical power is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No